CLINICAL TRIAL: NCT03662061
Title: Analysis of the Specific Onco-geriatric Multidisciplinary Team Meeting (RCP) at E.Herriot Hospital (Hospices Civils de Lyon)
Brief Title: Assessment of a Multidisciplinary Team Meeting (RCP) in Geriatric Oncology
Acronym: EROG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0674
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of the follow-up of oncological and geriatric recommendations 4 months after the RCP — After inclusion, patient's results are discussed at a weekly onco-geriatric multidisciplinary team meeting including surgeons, geriatrics, oncologists, radiotherapist, nurse, pharmacist. Oncological and geriatric recommendations are given.
  A phone call is made to the patient to evaluate the follow-up of the oncological and geriatric recommendations defined during the RCP along with their survival, autonomy and quality of life.

SUMMARY:
In France, cancer incidence increases over the course of life and therefore it is considered as an important pathology of the elderly. Cancers are the second leading cause of death for patients over 70 years old.

In 2015, 233,343 new cases of cancer were estimated for patients of 65 years and over (60.9% of estimated cancers of all ages), 42,547 new cases for older people over 85 years old (about 11% of all diagnosed cancer cases).

With the expected aging of the population in the coming years, the number of patients over the age of 70 will continue to increase. Life expectancy will also increase (12 years for the people above 75 years old and more than 8 years for the people above 80 years old).

The elderly are a heterogeneous population. Some people age well with few chronic diseases and a preserved autonomy. Others have several pathologies, geriatric syndromes (malnutrition, functional disorders, sensory deficits or psycho-cognitive diseases). Poly-medication is therefore common with an increased risk of iatrogenic disease. All these factors, in addition to social and economic conditions, determine the health status of the elderly. The presence of comorbidities decreases life expectancy and may itself be a contraindication to treatment. Patients in this age group are therefore particularly exposed to the risks of over- or under-treatment.

The multidisciplinary team meeting (RCP) is widely used for decision making in oncology. Various official texts govern it (Plan Cancer, HAS). However, the onco-geriatric decision is usually only a complementary opinion after a RCP of a specific organ.

Since 2006, the E. Herriot Hospital's Multidisciplinary team meeting has been organized to discuss cases of patients over 70 years old. The specificity is the association of a real multidisciplinary geriatric oncology discussion. The latter between medical specialist : geriatrician, oncologist, surgeon, radiotherapist, pharmacist, onco-geriatric nurse allows the development of an appropriate individualized therapeutic project for the patient.

The onco-geriatric multidisciplinary team is implementing a descriptive study of the RCP for the management of patients above 70 with cancer. The Regional Network of Oncology Auvergne-Rhône-Alpes is a partner.

The main aim is to describe the feasibility of the assessment of the follow-up of onco-geriatric recommendations 4 months after the onco-geriatric RCP of E. Herriot Hospital concerning patients with or with suspicion of cancer.

The secondary aims are : 1/ To describe the process of RCP: participants, patient's characteristics and conclusions with recommendations, 2/ To assess the implementation of oncological and geriatric recommendations 4 months after RCP 3/ To assess the survival, autonomy and quality of life of patients 4 months after RCP.

The hypothesis is that onco-geriatric RCP's recommendations improve the outcome for the patient.

The purpose of this pilot study is to ensure that the assessment of the recommendations' follow-up at 4 months is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years
* with cancer or suspicion of cancer,
* with a systematic collection of oncological and geriatric data in their medical record submitted to the onco-geriatric RCP of E. Herriot hospital.
* Patients must be able to express their non-opposition to participate in this study or must be accompanied by a trustworthy person able to express his or her opposition.

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study concerns patients above 70 years with cancer or suspicion of cancer who benefit from an onco-geriatric case analysis by the multidisciplinary team meeting (RCP).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose recommendations' follow-up at 4 months after RCP, has been feasible. | 4 months
  Phone call 4 months after RCP to assess if recommendations have been followed.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Oncologie radiothérapie - Hôpital Privé Jean Mermoz Ramsay Général de Santé Lyon, Lyon
  - Médecine Gériatrique/équipe mobile de gériatrie - Hôpital Edouard Herriot, Lyon

IPD SHARING:
Plan to Share IPD: No